CLINICAL TRIAL: NCT02939898
Title: Reducing the Impact of Ovarian Stimulation - The RIOT Project Study RIOT-B: Mapping the Endocrine Determinants of Ovarian Stimulation to Optimize Outcomes in Fresh Embryo Transfer Cycles
Brief Title: Mapping the Endocrine Determinants of Ovarian Stimulation to Optimize Outcomes in Fresh Embryo Transfer Cycles
Acronym: RIOT-B
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sven O. Skouby (Other)
Collaborators: Rigshospitalet, Denmark (Other); Region Capital Denmark (Other); Copenhagen University Hospital, Denmark (Other)
Responsible Party: Sponsor-Investigator, Sven O. Skouby, Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIOTB2015; 2015-005683-41 (EudraCT Number); H-15021852 (Other: Ethics Committee); HGH-2016-033_I-Suite: 04482 (Other: Danish Data Protection Board)
Record Dates: First submitted 2016-08-15; First posted 2016-10-20 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Letrozole; Aromatase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactose Monohydrate (Placebo Comparator): 2 tablets of placebo are administered daily from stimulation start to day before hCG as adjunctive therapy to 150 International Units of recFSH
  Interventions: Drug: Placebo
- Letrozole (Active Comparator): 2 tablets of 2,5 mg Letrozole are administered daily from stimulation start to day before hCG as adjunctive therapy to 150 International Units of recFSH
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Placebo — Adjuvant therapy to recFSH during ovarian stimulation
  Other Names: Lactose Monohydrate
  Arms: Lactose Monohydrate
Drug: Letrozole — Adjuvant therapy to recFSH during ovarian stimulation
  Other Names: Aromatase Inhibitor
  Arms: Letrozole

SUMMARY:
The goal of this project is to identify autocrine, paracrine and endocrine factors which are associated with intercycle variation in cyclical follicle recruitment.

Patients will be monitored in a natural cycle, a stimulated cycle and a follow up. In the stimulated cycle patients will be randomized to co-treatment with aromatase inhibitor or placebo during ovarian stimulation.

DETAILED DESCRIPTION:
The primary aim of this project is to explore the putative cyclic recruitment 'gatekeeping' functions of gonadotropins, sex steroids, anti-muellarian hormone and pregnancy associated plasma protein A in normal ovulatory cycles, and the impact of ovarian stimulation on cyclic follicle recruitment in the following cycle.

It is further proposed that supra-physiological levels of estradiol and progesterone which arise from ovarian stimulation may modulate the size of the secondarily recruited follicle cohort in the next cycle. In order to explore the relative contribution of sex steroids as determinants of the size of the next cycle 'wave' of recruitment further, a second aim of this study will be investigate whether limiting the rise in sex steroid levels during ovarian stimulation, by co-treatment with aromatase inhibitor impacts on cyclic recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Indication for IVF/ICSI treatment
* Eligible for IVF/ICSI treatment according to local criteria
* Regular cycles 21-35 days (both included)
* Age <40 years
* AMH 8-32 (both included)
* Written consent
* Willing to undergo intensive monitoring in a natural cycle (the cycle prior to the monitored natural cycle must be hormone treatment free), stimulated cycle and follow up in the subsequent cycle

Exclusion Criteria:

* Any contraindication for IVF/ICSI treatment according to local criteria
* Previous stimulation for IVF/ICSI with < 4 oocytes obtained
* PCOS
* Undergoing IVF/ICSI for the purpose of fertility preservation
* Allergy towards study drug

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Size of follicle cohort in relation to serum endocrine and paracrine markers | The change in size of follicle cohort in relation to change in endocrine and paracrine markers assessed throughout the study completion, up to 3 years.
  Markers for analysis include: anti-muellerian hormone, estradiol, follicle stimulating hormone, luteinizing hormone, testosterone, androstenedione, progesterone,17-hydroxyprogesterone, pregnancy associated plasma protein A and A2, Inhibin A and B, Bone morphogenic protein

SECONDARY OUTCOMES:
Size of the cyclically recruited follicle cohort after ovarian stimulation with and without co-treatment with Aromatase Inhibitor. | The change in size of follicle cohort throughout the study completion, up to 3 years.
Expression of cytokine and growth factors in endometrial secretions following co-treatment with Aromatase Inhibitor compared with placebo control. | Assessed in stimulated cycle at time of embryo transfer (throughout study completion, up to 3 years).
Serum E2, P, Tst and Androstenedione levels | The change in levels throughout the study completion, up to 3 years.
Area under the curve for P and 17-hydroxyprogesterone. | The change in levels throughout the study completion, up to 3 years.
Total International Units of Follicle Stimulating Hormone used per treatment cycle. | Assessed throughout study completion, up to 3 years.
Number of follicles > 12 mm | Assessed throughout the study completion, up to 3 years.
Number of oocytes obtained | Assessed during stimulation treatment (throughout the study completion, up to 3 years).
Proportion of oocytes resulting in top quality day 2, day 3 embryos or day 5/6 embryos according to validated morphological criteria. | Assessed during stimulation treatment (throughout the study completion, up to 3 years).
Oocyte fertilization rate | Assessed during stimulation treatment (throughout the study completion, up to 3 years).
Number and quality of embryos obtained. | Assessed during stimulation treatment (throughout the study completion, up to 3 years).
Endometrial thickness | Assessed throughout the study completion, up to 3 years.
Uterine contraction rate (contractions/minute) | Assessed throughout the study completion, up to 3 years.
Implantation rate | Assessed during stimulation treatment (throughout the study completion, up to 3 years).
Reported side effects | From start of stimulation and administration of study medication to pregnancy scan week gestational age 7-8. Assessed throughout the study completion, up to 3 years.
Morphokinetic parameters of embryo quality as measured using a Time Lapse analysis. | Assessed from time of oocyte pick-up to embryo transfer following stimulation (throughout study completion, up to 3 years)
Clinical pregnancy rate | Pregnancy scan at gestational age week 7-8 (3-4 weeks after the positive hCG in serum) Assessed during stimulation treatment (throughout the study completion, up to 3 years).
Follicular fluid endocrine and paracrine markers following co-treatment with Aromatase Inhibitor compared with placebo control. | Assessed during stimulation treatment (throughout the study completion, up to 3 years).
Biochemical pregnancy rate | Assessed during stimulation treatment (throughout the study completion, up to 3 years).
Area under the curve for E2, P and LH | The change in levels throughout the study completion, up to 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Sven O. Skouby, Professor, Principal Investigator — Unit of Reproductive Medicine, Herlev/Gentofte Hospital
Locations (1):
- Unit of Reproductive Medicine, Herlev Hospital, Herlev, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The study will share data with Study RIOT-A

REFERENCES:
- [Derived] Bulow NS, Warzecha AK, Nielsen MV, Andersen CY, Holt MD, Petersen MR, Sopa N, Zedeler A, Englund AL, Pinborg A, Grondahl ML, Skouby SO, Macklon NS. Impact of letrozole co-treatment during ovarian stimulation on oocyte yield, embryo development, and live birth rate in women with normal ovarian reserve: secondary outcomes from the RIOT trial. Hum Reprod. 2023 Nov 2;38(11):2154-2165. doi: 10.1093/humrep/dead182. PMID 37699851
- [Derived] Poulsen LC, Warzecha AK, Bulow NS, Bungum L, Macklon NS, Yding Andersen C, Skouby SO. Effects of letrozole cotreatment on endocrinology and follicle development in women undergoing ovarian stimulation in an antagonist protocol. Hum Reprod. 2022 Jun 30;37(7):1557-1571. doi: 10.1093/humrep/deac119. PMID 35652260
- [Derived] Dreyer Holt M, Warzecha AK, Bulow NS, Skouby SO, Englund ALM, Birch Petersen K, Macklon NS. Does adjuvant letrozole reduce uterine peristalsis prior to fresh embryo transfer? Hum Reprod Open. 2022 Mar 8;2022(2):hoac011. doi: 10.1093/hropen/hoac011. eCollection 2022. PMID 35356508
- [Derived] Bulow NS, Skouby SO, Warzecha AK, Udengaard H, Andersen CY, Holt MD, Grondahl ML, Nyboe Andersen A, Sopa N, Mikkelsen ALE, Pinborg A, Macklon NS. Impact of letrozole co-treatment during ovarian stimulation with gonadotrophins for IVF: a multicentre, randomized, double-blinded placebo-controlled trial. Hum Reprod. 2022 Jan 28;37(2):309-321. doi: 10.1093/humrep/deab249. PMID 34792133